CLINICAL TRIAL: NCT03412253
Title: From Diabetes Care to Diabetes Cure; Could Single-anastomosis Gastric Bypass Be a Safe Bridge to Reach This Target in Non-Obese Patients?
Brief Title: Could Single-anastomosis Gastric Bypass Be a Curative Treatment for Type II Diabetes?
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: financial causes, and the study will be continued within days.
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Tarek Abouzeid Osman Abouzeid, Principal Investigator, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1349
Record Dates: First submitted 2018-01-13; First posted 2018-01-26 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Metabolic Surgery
Keywords: metabolic surgery, BMI 25-30 kg/m2, SAGB, T2DM remission.

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Single-Anastomosis Gastric Bypass surgery (SAGB). — We checked the effect of SAGB on patients suffered from T2DM with BMI 25-30
  Other Names: Mini-Gastric Bypass.; One-Anastomosis Gastric Bypass.

SUMMARY:
Single- Anastomosis gastric bypass (SAGB) is a potentially curative line of treatment for type II diabetes mellitus (T2DM) patients with BMI 25-30 kg/m2. Accordingly, SAGB could be integrated into T2DM treatment algorithm

DETAILED DESCRIPTION:
Background: T2DM has been considered as a chronic progressive incurable metabolic disease. Single-anastomosis gastric bypass (SAGB) was shown to be effective in obese patients in terms of weight reduction and T2DM remission, yet its effect on non-obese diabetics is not extensively studied. In this study, we tried to determine the anthropometric and glycemic outcomes of SAGB as a proposed line of treatment for type II diabetes mellitus (T2DM) patients with body mass index (BMI) 25-30 kg/m2.

Methods: From November 2013 to March 2016, a prospective study has been conducted at Ain-Shams University hospitals on 17 consecutive patients undergone SAGB. The demographic and anthropometric data of the patients, as well as their relevant laboratory results, were reported, other data including anti-diabetic medications, co-morbid metabolic diseases were also assessed. All patients were scheduled for laparoscopic SAGB and were advised to come in regular follow up at 1, 3, 6, 12 and 18 months postoperatively. T2DM Remission is considered if glycosylated hemoglobin (HbA1c) <6.5 % and fasting plasma glucose (FPG) < 126 mg/dl for at least 1 year without medication.

ELIGIBILITY:
Inclusion Criteria:

.Type II diabetic patients.

* Age: 20-60 years.
* either gender.

Exclusion Criteria:

* Previous bariatric surgery.
* Controlled T2DM.
* Duration of T2DM >10 years.
* Patients with endocrinal diseases,
* Pregnancy.
* Those unfit for general anesthesia.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2018-02-04 (Estimated)

PRIMARY OUTCOMES:
Cure of type II DM. | 1Year
  T2DM Remission is considered if glycosylated hemoglobin (HbA1c) <6.5 % and fasting plasma glucose (FPG) < 126 mg/dl for at least 1 year without medication.

IPD SHARING:
Plan to Share IPD: Undecided